CLINICAL TRIAL: NCT06280768
Title: A Phase Ib Clinical Study to Evaluate the Safety and Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Subcutaneous Injections of SHR-2004 Injection in Patients With Atrial Fibrillation
Brief Title: Study on the Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of SHR-2004 Injection in Adult Patients With Atrial Fibrillation
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Suncadia Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-2004-102
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-2004 injection (Experimental)
  Interventions: Drug: SHR-2004 injection

INTERVENTIONS:
Drug: SHR-2004 injection — dose 1 or dose 2 or dose 3 or dose 4 or dose 5 or dose 6

SUMMARY:
This study is an open-label Phase Ib clinical study with the primary objective of evaluating the safety and tolerability of multiple subcutaneous injections of SHR-2004 injection in patients with atrial fibrillation, and the secondary objective is to evaluate its pharmacokinetic (PK), pharmacodynamic (PD) and immunogenicity characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the study procedures and methods, voluntarily participate in this trial, and sign the informed consent form in writing;
2. Male or female ≥ 40 years and < 80 years old；
3. History of atrial fibrillation or atrial flutter, or newly diagnosed atrial fibrillation or atrial flutter during the screening period, as documented by Holter ECG or 12-lead ECG at the time of screening or within 12 months prior to screening.

Exclusion Criteria:

1. Patients with a mechanical heart valve;
2. Rheumatic mitral stenosis or moderate to severe non-rheumatic mitral stenosis;
3. Atrial fibrillation or atrial flutter is caused by reversible causes, or successful ablation has been converted to sinus rhythm, or cardioversion or ablation surgery is planned during the study;
4. Concomitant poorly controlled hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100mmHg) at screening;
5. Those who are allergic to the trial drug or any component of the trial drug;
6. Unstable or severe liver, renal, cardiovascular, psychiatric, neurological, endocrine, hematological and other diseases at the time of screening, and the investigator judges that it is not suitable to participate in the study;
7. Females who are pregnant or lactating.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (including bleeding events) | Up to 136 Days

SECONDARY OUTCOMES:
Pharmacokinetics of SHR2004: Peak Plasma Concentration (Cmax) | Up to 136 Days
Pharmacokinetics of SHR2004: Area under the plasma concentration versus time curve (AUC) | Up to 136 Days
Pharmacokinetics of Dupilumab: Elimination half life (t1/2) | Up to 136 Days
PD endpoint: absolute and relative change values of coagulation factor XI (FXI) activity | Up to 136 Days
PD endpoint: absolute and relative change values of activated partial thromboplastin time (APTT) | Up to 136 Days
Immunogenicity endpoint: the incidence and timing of ADA positivity in SHR-2004 | Up to 136 Days

IPD SHARING:
Plan to Share IPD: Undecided